CLINICAL TRIAL: NCT05045196
Title: Health-promoting Family Conversations and Open Heart Surgery -An Intervention Model for Families: The HeartFam Intervention
Brief Title: Health-promoting Family Conversations and Open Heart Surgery
Acronym: HeartFam
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Örebro University, Sweden (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 4.2-05418/2020
Record Dates: First submitted 2020-11-13; First posted 2021-09-16 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Thoracic Surgery
Keywords: Family Nursing

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient and family member of patient undergoing elective open heart surgery- Intervention (Experimental): Family randomized to the intervention group receiving Health-promoting conversation intervention
  Interventions: Behavioral: Health promoting conversations
- Patient and family member of patient undergoing elective open heart surgery- Control (No Intervention): Family of a patient undergoing elective open-heart surgery randomized to the intervention group receiving standard care

INTERVENTIONS:
Behavioral: Health promoting conversations — The Health-promoting conversations intervention is a conversation model between the patient, family members, and a trained nurse. Patients and families included in the study will, after submitting base-line-data, be randomized to
  Arms: Patient and family member of patient undergoing elective open heart surgery- Intervention

SUMMARY:
Elective open-heart surgery involves physical and psychological strain for the person undergoing surgery. Family plays a significant part in care before and after surgery, and the family has care needs of their own. Health services need to address the family-caregiver burden as an essential aspect of care. Different methods aiming at stress reduction and involvement of patients and family members in care exist. The evidence is conflicting concerning which way is the most effective. Health-promoting conversations are an intervention model promoting family well-being and alleviation of illness and illness-related suffering for the whole family.

Families´ in the intervention group in this trial will, before and after one family member's elective open-heart surgery, participate in Health-promoting conversations. Health-promoting conversation is an intervention model based on the Family Systems Nursing theory. The person undergoing surgery decides which family members should be asked to participate in 1-3 conversations whit a family nurse. Effects on postoperative recovery, health-related quality of life, stress, and patient and family involvement in care will be evaluated with patient- and family-reported outcome measures.

The aim is to evaluate Health-promoting conversation's effect on family wellbeing, functioning, and involvement in care. The cost-effectiveness of the intervention will also be evaluated.

The study will follow the ethical guidelines of the Declaration of Helsinki. The Swedish National Committee on Health Research Ethics reviewed and accepted the study in march 2020 (nr 2019-06315)

ELIGIBILITY:
Inclusion Criteria

Patients:

* Patients =/>18 years of age
* undergoing elective, open-heart surgery
* having a minimum of one family member willing to participate in Health-promoting conversations

Family members

* Family member of a patient undergoing elective, open-heart surgery
* willing to participate in Health-promoting conversations *=/> 15 years of age

Exclusion Criteria patient and family member:

* Inability to speak or understand Swedish to the extent of giving informed consent
* Cognitive and/or psychiatric disorder to the extent of not being able to give informed consent

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 267 (Actual)
Dates: Start 2022-09-16 (Actual); Primary Completion 2024-06-02 (Actual); Study Completion 2025-03-15 (Actual)

PRIMARY OUTCOMES:
Family-Sense Of Coherence (F-SOC) | A statistically significant change in F-SOC from baseline at three months after hospital discharge between the trial patient groups.
  Person-reported outcome measure, questionnaire measuring sense of coherence at family level. 12 items.

SECONDARY OUTCOMES:
RAND-36 | Baseline (before randomization)
  Swedish version of Short Form-36 (SF-36) a questionnaire measuring health-related quality of life. 36 items, 8 dimensions.
RAND-36 | 2 weeks after hospital discharge
  Swedish version of Short Form-36 (SF-36) a questionnaire measuring health-related quality of life. 36 items, 8 dimensions.
RAND-36 | 3 month follow up
  Swedish version of Short Form-36 (SF-36) a questionnaire measuring health-related quality of life. 36 items, 8 dimensions.
RAND-36 | 12 month follow up
  Swedish version of Short Form-36 (SF-36) a questionnaire measuring health-related quality of life. 36 items, 8 dimensions.
Family Involvement in Care Questionnaire (FICQ) | Family members only: 2 weeks after hospital discharge
  Person-reported outcome measure, questionnaire measuring family members perceived Instrument measuring family members experiences of involvement in care of the family member who is a patient. 16 items on a 4-point Likert-scale and 2 open ended questions.
Cost-Effectiveness of Heath promoting conversations | Baseline (before randomization)
  A questionnaire measuring care utilization and absence from work, 12 items.
Cost-Effectiveness of Heath promoting conversations | 2 weeks after hospital discharge
  A questionnaire measuring care utilization and absence from work, 12 items.
Cost-Effectiveness of Heath promoting conversations | 3 month follow up
  A questionnaire measuring care utilization and absence from work, 12 items.
Cost-Effectiveness of Heath promoting conversations | 6 month follow up
  A questionnaire measuring care utilization and absence from work, 12 items.
Cost-Effectiveness of Heath promoting conversations | 12 month follow up
  A questionnaire measuring care utilization and absence from work, 12 items.
Postoperative Recovery Profile (PRP) | Baseline
  Person-reported outcome measure, questionnaire measuring self-reported postoperative recovery. 19 items, 5 dimensions and a cardiac surgery specific module consisting of 7 items at baseline.
Postoperative Recovery Profile (PRP) | 2 weeks after hospital discharge
  Person-reported outcome measure, questionnaire measuring self-reported postoperative recovery. 19 items, 5 dimensions and a cardiac surgery specific module consisting of 9 items.
Postoperative Recovery Profile (PRP) | 3 month follow up
  Person-reported outcome measure, questionnaire measuring self-reported postoperative recovery. 19 items, 5 dimensions and a cardiac surgery specific module consisting of 9 items.
Postoperative Recovery Profile (PRP) | 12 month follow up
  Person-reported outcome measure, questionnaire measuring self-reported postoperative recovery. 19 items, 5 dimensions and a cardiac surgery specific module consisting of 9 items.
Family-Sense Of Coherence (F-SOC) | Baseline (before randomization)
  Person-reported outcome measure, questionnaire measuring sense of coherence at family level. 12 items.
Family-Sense Of Coherence (F-SOC) | 2 weeks after hospital discharge
  Person-reported outcome measure, questionnaire measuring sense of coherence at family level. 12 items.
Family-Sense Of Coherence (F-SOC) | 12 month follow up
  Person-reported outcome measure, questionnaire measuring sense of coherence at family level. 12 items.
Family Hardiness Index (FHI) | Baseline
  Measurement of the persons perceived hardiness within the family, consisting of 20 items on a 4-point Likert scale.
Family Hardiness Index (FHI) | 2 weeks after hospital discharge
  Measurement of the persons perceived hardiness within the family, consisting of 20 items on a 4-point Likert scale.
Family Hardiness Index (FHI) | 3 month follow up
  Measurement of the persons perceived hardiness within the family, consisting of 20 items on a 4-point Likert scale.
Family Hardiness Index (FHI) | 12 month follow up
  Measurement of the persons perceived hardiness within the family, consisting of 20 items on a 4-point Likert scale.
General Functioning Scale (GFS) | Baseline
  Measurement of the persons perceived family functioning, 12 items on a 4-point Likert scale.
General Functioning Scale (GFS) | 2 weeks after hospital discharge
  Measurement of the persons perceived family functioning, 12 items on a 4-point Likert scale.
General Functioning Scale (GFS) | 3 month follow up
  Measurement of the persons perceived family functioning, 12 items on a 4-point Likert scale.
General Functioning Scale (GFS) | 12 month follow up
  Measurement of the persons perceived family functioning, 12 items on a 4-point Likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Ericsson, Principal Investigator — Örebro University, Sweden
Locations (3):
- Sweden (3):
  - Department of Cardiovascular and Thoracic Surgery, Örebro University Hospital, Örebro, Närke
  - Thoracic Surgery and Anesthesia, Uppsala university hospital, Uppsala, Uppland
  - Department of Thoracic and Vascular Surgery Linköping university hospital, Linköping, Östergötland County